CLINICAL TRIAL: NCT02696629
Title: The Impact of Sleep Apnea Treatment on Physiology Traits in Chinese Patients With Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, YANRU LI, M.D., Beijing Tongren Hospital
Other Study IDs: TRECKY2013-004-1
Record Dates: First submitted 2016-02-26; First posted 2016-03-02 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: Ventilatory control; Obstructive sleep apnea; Loop gain; Upper airway; Surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Education and follow up: Participants who refuse or fail to have PAP treatment or Oral appliance or other treatments for sleep apnea. They also refuse or have counter-indication for surgical treatment. The impact of weight loss, sleep position, alcohol avoidance, risk factor modification and medication effects and follow-up are provided for patients' education.
  Interventions: Behavioral: education and follow up
- Upper airway surgery: Participants who undergo uvulopalatopharyngoplasty, concomitant transpalatal advancement pharyngoplasty, nasal surgery or multi-level upper airway surgery.
  Interventions: Procedure: upper airway surgery
- Continues positive airway pressure: Participants who are treated with continues positive airway pressure during sleep.
  Interventions: Device: Continues positive airway pressure

INTERVENTIONS:
Procedure: upper airway surgery — Uvulopalatopharyngoplasty, concomitant transpalatal advancement pharyngoplasty, nasal surgery or multi-level upper airway surgery
  Groups: Upper airway surgery
Device: Continues positive airway pressure — Participants who are treated with continues positive airway pressure during sleep.
  Groups: Continues positive airway pressure
Behavioral: education and follow up — Patients education and follow up:The impact of weight loss, sleep position, alcohol avoidance, risk factor modification and medication effects and follow-up are provided for patients' education.
  Groups: Education and follow up

SUMMARY:
The prevalence of OSA is 3.5~4.6% in Chinese adults. OSA leads to repetitive hypoxemia, hypercapnia, and arousal from sleep and is an independent risk factor for hypertension, stroke, coronary artery disease and congestive heart failure. CPAP is the first-line treatment for OSA. But many patients do not adhere to therapy.

The upper airway(UA) anatomical abnormality is a prominent risk factor in Asian OSA patients, which might be improved by surgical strategies. However, surgery shows variable clinical effectiveness. One important reason for patients responding poorly to single treatment procedure is that multiple abnormal physiological traits contribute to OSA.

High loop gain is one of the key non-anatomical risk factors. It will be useful to individualize therapy in OSA by better understanding the reversibility of increased LG, the interaction of LG and UA anatomical change as well as the condition that trigger reduction of LG.

The project will test the hypothesis of 1) Elevated LG is induced in some patients and is reversible by treatment of OSA; 2) Change of LG is related to the improvement of sleep apnea; 3) An elevated LG is related to residual sleep apnea after upper airway surgery, which might be eliminated by adjunct CPAP therapy after surgery. The results would improve the efficiency of non-CPAP treatment and provide a potential combined treatment option for those patients with both elevated loop gain and anatomy risk factors in the Asian population.

DETAILED DESCRIPTION:
Unstable respiratory control (high loop gain) is an important non-anatomical risk factor for obstructive sleep apnea. Studies showed high loop gain might also be acquired from long-term hypoxemia/hypercapnia due to OSA, and could be decreased by CPAP therapy in some of the individuals. Whether another treatment, i.e. upper airway surgery, could achieve a similar improvement in is not known. We hypothesize that 1) high LG could be reversible with improved hypoxemia and reduced apnea hypopnea index (AHI) by surgical treatment; 2) high loop gain at baseline may be associated with poor treatment outcomes.

PSG was performed pre- and postoperatively to assess the OSA severity in participants who underwent uvulopalatopharyngoplasty and concomitant transpalatal advancement pharyngoplasty. Loop gain were calculated using a published method by fitting a feedback control model to airflow. The loop gain values at baseline and follow-up were compared. The association between loop gain change and improvement of OSA were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70 years
* Sleep study (with apnea-hypopnea index>5)
* Diagnosis of obstructive sleep apnea

Exclusion Criteria:

* Any known unstable cardiac (apart from treated hypertension), pulmonary, renal, neurologic (including epilepsy), thyroid, neuromuscular, or hepatic disease
* Pregnant women or nursing mothers
* Use of any medications that may affect sleep or breathing
* An uncontrolled psychiatric disorder
* Use of illicit drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obstructive sleep apnea
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-11 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in ventilatory control after intervention | 6 month to 1 year
  Loop gain at a disturbance of frequency 1 cycle/minute were calculated using a published method by fitting a feedback control model to airflow
Change from baseline in sleep apnea severity after intervention | 6 month to 1 year
  Assess using standard sleep scoring criteria

SECONDARY OUTCOMES:
Change from baseline in upper airway anatomy after surgery | 6 month to 1 year
  Upper airway computed tomography
Change from baseline in symptoms after intervention | 6 month to 1 year
  Assess using questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Demin Han, M.D, Ph.D, Study Director — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wellman A, Jordan AS, Malhotra A, Fogel RB, Katz ES, Schory K, Edwards JK, White DP. Ventilatory control and airway anatomy in obstructive sleep apnea. Am J Respir Crit Care Med. 2004 Dec 1;170(11):1225-32. doi: 10.1164/rccm.200404-510OC. Epub 2004 Aug 18. PMID 15317668
- [Background] Owens RL, Edwards BA, Eckert DJ, Jordan AS, Sands SA, Malhotra A, White DP, Loring SH, Butler JP, Wellman A. An Integrative Model of Physiological Traits Can be Used to Predict Obstructive Sleep Apnea and Response to Non Positive Airway Pressure Therapy. Sleep. 2015 Jun 1;38(6):961-70. doi: 10.5665/sleep.4750. PMID 25515107
- [Background] Terrill PI, Edwards BA, Nemati S, Butler JP, Owens RL, Eckert DJ, White DP, Malhotra A, Wellman A, Sands SA. Quantifying the ventilatory control contribution to sleep apnoea using polysomnography. Eur Respir J. 2015 Feb;45(2):408-18. doi: 10.1183/09031936.00062914. Epub 2014 Oct 16. PMID 25323235
- [Background] Loewen A, Ostrowski M, Laprairie J, Atkar R, Gnitecki J, Hanly P, Younes M. Determinants of ventilatory instability in obstructive sleep apnea: inherent or acquired? Sleep. 2009 Oct;32(10):1355-65. doi: 10.1093/sleep/32.10.1355. PMID 19848364
- [Derived] Li Y, Ye J, Han D, Zhao D, Cao X, Orr J, Jen R, Deacon-Diaz N, Sands SA, Owens R, Malhotra A. The Effect of Upper Airway Surgery on Loop Gain in Obstructive Sleep Apnea. J Clin Sleep Med. 2019 Jun 15;15(6):907-913. doi: 10.5664/jcsm.7848. PMID 31138381
- [Derived] Li Y, Ye J, Han D, Cao X, Ding X, Zhang Y, Xu W, Orr J, Jen R, Sands S, Malhotra A, Owens R. Physiology-Based Modeling May Predict Surgical Treatment Outcome for Obstructive Sleep Apnea. J Clin Sleep Med. 2017 Sep 15;13(9):1029-1037. doi: 10.5664/jcsm.6716. PMID 28818154